CLINICAL TRIAL: NCT01219647
Title: Exercise as a Strategy to Treat Cognitive Dysfunction in Persons With Multiple Sclerosis
Acronym: CogEx
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: California State University, Northridge (Other)
Responsible Party: Principal Investigator, Barbara Giesser, Clincial Profesor of Neurology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RG 4174A5/2
Record Dates: First submitted 2010-10-08; First posted 2010-10-13 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Exercise; Cognition
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- aerobic exercise (Experimental): Subjects will train on a recumbent cross trainer 20-30 minutes/session for three times/week for six months under supervision of a fitness specialist
  Interventions: Behavioral: exercise
- stretching (Active Comparator): Subjects will particiate in supervised stretching at same frauency, duration and intensity of aerobic exericse arm
  Interventions: Behavioral: stretching

INTERVENTIONS:
Behavioral: exercise — subjects will participate in one of two forms of exercise
  Arms: aerobic exercise
Behavioral: stretching — subjects will particiopate in supervised stretching as described in arm description.
  Arms: stretching

SUMMARY:
Many persons with Multiple Sclerosis ( MS) have problems with memory and thinking.Exercise has been shown to improve memory and thinking in persons with diseases such as Alzheimer's. This study will investigate whether a program of aerobic exercise can improve memory and thinking in persons with MS

DETAILED DESCRIPTION:
Persons with Multiple Sclerosis(MS)will be screened for eligibility and randomized to a protocol with two intervention arms. One group will have aerobic training on a recumbent cross trainer three times a week for 20-30 minutes/session. The other group will participate in stretching exercises at the same frequency and intensity.Total training time will be six months.Outcome measures will include tests of memory and thinking, and fitness measures.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of MS Complaints of cognitive problems Able to ride a recumbent cross trainer

Exclusion Criteria:

* Cardiopulmonary or structural disease that would limit ability to participate in exercise training On treatment with chemotherapy or natalizumab Screening score of >50 on PASAT

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2010-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Paced Auditory Serial Addition Test (PASAT) | 36 weeks
  test of attention and information processing

SECONDARY OUTCOMES:
Symbol Digit Modalities Test (SDMT) | 36 weeks
  test of attention and information processing
VO2 max | 36 weeks
  measure of fitness via oxygen consumption and use
Long latency cognitive event related potentials ( LLCERP) | 36 weeks
  electrophysiologic tests of information processing

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Giesser, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - UCalifornia at Los Angeles, Los Angeles, California
  - CAl State University at Northridge, Northridge, California